

## $\underline{\textbf{P}} \textbf{ati} \underline{\textbf{E}} \textbf{nt} \ \underline{\textbf{N}} \textbf{europsychological outcome} \underline{\textbf{S}} \ \underline{\textbf{A}} \textbf{fter lase} \underline{\textbf{R}} \ \textbf{ablation}$



Statistical Plan August 21, 2021 Study objectives will not be statistically powered given the anticipated heterogeneity in available neuropsychological test results.

Scores will be collected to assess domain specific changes for the Primary outcome measure using pre-defined clinically meaningful cut scores (based on previously described methods):

- Changes of 1.5 standard deviations will be considered improved (+) or worsened (-).
- Changes of 2.5 standard deviations will be considered substantial post-operative improvements (+) or worsening (-).
- Any score change less than 1.5 standard deviation will be considered unchanged and the result of anticipated variability.

Descriptive statistics will be used to summarize the results for Secondary Outcome measures:

- Continuous variables: The total count, mean, standard deviation, minimum, and maximum will be provided.
- Categorical variables: Total count and percentage will be provided.

Ad hoc, exploratory analyses may be conducted if sufficient sample size allows for correlation or multivariate assessment of patient subsets (e.g., those with improvement or worsening).